CLINICAL TRIAL: NCT06785883
Title: Screening Anxiety and Depression Among Patients with Chronic Musculoskeletal Pain Within Physiotherapy Practices
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Davy Vancampfort, Professor, KU Leuven
Other Study IDs: S67100
Record Dates: First submitted 2025-01-03; First posted 2025-01-21 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2025-01

CONDITIONS: Osteoarthitis; Fibromyalgia; Rheumatoid Arthritis (RA; Low Back Pain; Neck Pain
MeSH Terms: conditions — Fibromyalgia; Arthritis, Rheumatoid; Low Back Pain; Neck Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study will investigate whether physiotherapists can accurately identify symptoms of anxiety and of depression in patients with chronic musculoskeletal pain (primary aim). The prevalence of co-morbid anxiety and depression in patients with chronic neck and / or shoulder pain, chronic low back pain, rheumatoid arthritis, osteoarthritis or fibromyalgia within physiotherapy practices will be established (secondary aim).

DETAILED DESCRIPTION:
The International Classification of Diseases describes chronic musculoskeletal pain as pain that arises as part of a disease process directly affecting bones, joints, muscle or related soft tissue lasting longer than 3 months. The global burden of chronic musculoskeletal pain is substantial, with a recent systematic review indicating a 26% prevalence in the general adult population and 39% in those older than 65 year. Chronic musculoskeletal pain also contributes to almost 20% of the global years-lived with disability, and it is one of the major causes of work loss and early retirement. Population-based research has shown that chronic pain conditions are risk factors for developing depression and anxiety. Co-morbid depression and anxiety are strongly associated with more severe pain, greater disability, and poorer health related quality of life. Both are also important reasons for poor treatment adherence within physiotherapy practices. When managing patients with chronic musculoskeletal pain, physiotherapists need to be able to identify patients who have an increased likelihood of depression and anxiety and to facilitate appropriate management by either facilitating patients in coping with anxiety and depression via for example physical activity or relaxation techniques and/or referring them to a medical practitioner for definitive diagnosis and intervention. Although there is some recognition of screening for depression in physiotherapy practices, the role physiotherapists can have in detecting anxiety and depression is largely ignored. The primary aim of this project will be to investigate whether physiotherapists can accurately identify symptoms of anxiety and of depression in patients with chronic musculoskeletal pain. The focus will in particular be on patients with chronic neck and / or shoulder pain, chronic low back pain, rheumatoid arthritis, osteoarthritis or fibromyalgia. The accuracy of screening via a numeric rating scale will be compared with the accuracy of screening via 2 brief items. A secondary aim is to describe the prevalence of co-morbid anxiety and depression in patients with chronic neck and / or shoulder pain, chronic low back pain, rheumatoid arthritis, osteoarthritis or fibromyalgia within physiotherapy practices.

ELIGIBILITY:
Inclusion criteria:

Physiotherapists:

- Physiotherapists of AXXON, the Belgian Professional Physiotherapy Organization.

Patients

- Self-reported chronic neck and / or shoulder pain, chronic low back pain, rheumatoid arthritis, osteoarthritis or fibromyalgia.

Exclusion criteria:

* Not meeting inclusion criteria.
* No additional exclusion criteria.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic pain
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-01-02 (Actual)

PRIMARY OUTCOMES:
Generalized Anxiety Disorder - 7 | 2 weeks
  The Generalized Anxiety Disorder Assessment (GAD-7) (14) is a seven-item instrument that is used to measure or assess the severity of anxiety symptoms. Each item asks the individual to rate the severity of their symptoms over the past two weeks. Each item is scored on a Likert scale with symptoms rated as 0 (not at all), 1 (several days), 2 (more than half the days) and 3 (nearly every day). The total score ranges from 0 to 21. Higher scores implicate more severe symptoms. The optimal cut-off scores for the presence of mild, moderately severe and severe depressive symptoms is 5≤9, 10≤14 and 15≤ respectively (14).
Patient Health Questionnaire -9 | 2 weeks
  Patient Health Questionnaire-9 (PHQ-9) The PHQ-9 is a nine-item depression scale (13). Each item asks the individual to rate the severity of their symptoms over the past two weeks. Each item is scored on a Likert scale with symptoms rated as 0 (not at all), 1 (several days), 2 (more than half the days) and 3 (nearly every day). The total score ranges from 0 to 27. Higher scores implicate more severe symptoms. The optimal cut-off scores for the presence of mild, moderate and severe depressive symptoms is 5≤9, 10≤19, and 20≤ respectively (13).
Numeric Rating Scale | 2 weeks
  Each physiotherapist will be requested to complete a patient evaluation form with a 0-to-10 numeric rating scale to rate whether the patient they just treated exhibited symptoms of anxiety and / or depression. Ratings will be allocated as 0 = "not at all depressed" and "not at all anxious"; 5 = "depressed" and "anxious" and 10 = "extremely depressed" and "extremely anxious".

CONTACTS AND LOCATIONS:
Locations (1):
- Private physiotherapy practices, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No